CLINICAL TRIAL: NCT05728008
Title: Retrospective Observational Comparison Study Between Ustekinumab and Tofacitinib as Third Line Therapy in a Multicenter Cohort of Patients With Refractory Ulcerative Colitis.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mariangela Allocca, Gastroenterologist, IRCCS San Raffaele
Other Study IDs: UST-TOFA3
Record Dates: First submitted 2023-01-30; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Ustekinumab; tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- subject treated with ustekinumab (anti-IL12-23): subjects treated with ustekinumab (anti-IL12-23) and have a follow-up at 24 +/- 4 weeks from the start of the third line therapy
  Interventions: Drug: Ustekinumab
- subject treated withtofacitinib (pan JAK inhibitor): subjects treated with tofacitinib (pan JAK inhibitor) and have a follow-up at 24 +/- 4 weeks from the start of the third line therapy.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Ustekinumab — a human monoclonal antibody to interleukin IL 12/23 p40. It is indicated in the treatment of adult patients with moderately to severely active UC. The induction phase consists of approximately 6 mg/kg intravenous dose administration. After the induction, the maintenance phase consists of a 90mg subcutaneous dose every 8 weeks.
  Groups: subject treated with ustekinumab (anti-IL12-23)
Drug: Tofacitinib — Jak inhibitor. It is indicated in the treatment of adult patients with moderately to severely active UC who have experienced inadequate response or have lost the response or who are intolerant to conventional therapy or to a biological agent. The induction phase consists of 10mg twice daily for 8 to 16 weeks. After the induction, the maintenance phase consists of 5mg x twice daily.
  Groups: subject treated withtofacitinib (pan JAK inhibitor)

SUMMARY:
Ulcerative colitis (UC) is a chronic remitting and relapsing inflammatory bowel disease. The pathogenesis is multifactorial, involving genetic predisposition, epithelial barrier defects, dysregulated immune responses, and environmental factors. It is diagnosed through colonoscopy and histological evidence of mucosal inflammation involving predominantly the rectum and potentially extending continuously up to the proximal segments of the colon. The patients affected present with severe abdominal pain, bloody diarrhea together with extraintestinal manifestations such as peripheral arthritis, pyoderma gangrenosum, erythema nodosum, ankylosing spondylitis and many others. The last 20 years have been profitable from the therapeutical point of view thanks to the advent of biological drugs which are derived from a living organism or its products including antibodies, interleukins and other molecules capable to target specific cellular pathways and to modulate different mechanisms such as blocking the actions of cytokines or white cells movement in the gut. More recently new promising alternatives seems to be the so-called small molecule drugs which are chemically derived low molecular weight compounds capable to enter the cell to regulate its functions and more generally biological processes like inflammation. In the last years, the therapeutic offer for ulcerative colitis patients has been enriched with the advent of biologics with different mechanism of action and very recently with the availability of the small molecules. Currently the available therapeutic options for ulcerative colitis include topic and systemic mesalazine, topic and systemic glucocorticoids, immunosuppressants (thiopurines), biological drugs (anti-tumor necrosis factor α (TNFα), inhibitor of α4β7 integrin, anti-IL12-23) and small molecules (JAK inhibitors). However, if on the one hand the therapeutical enrichment has clearly improved the disease rate control, still there is the need to perform sequencing study to stratify the available options to provide the best and most appropriate patient-oriented management.

DETAILED DESCRIPTION:
This is an observational, retrospective, international multicenter study on the comparison of ustekinumab (anti-IL12-23) and tofacitinib (pan JAK inhibitor) used as third-line therapy in UC cases.

The aim of this retrospective multicentric observational study is to determine which between ustekinumab (anti-IL12-23) and tofacitinib (pan JAK inhibitor) as third-line therapy in UC cases refractory to both anti-TNFα and vedolizumab (inhibitor of α4β7 integrin) is the best compound to achieve disease control. The primary goal is to compare the hospitalization rate, surgery rate, drug optimization rate and the drug discontinuation rate, as a composite primary objective, in patients on either of the two drugs.

Subjects received the drugs, as per clinical practice, starting from their marketing authorization up to February 2022. The data will be collected starting from the time of diagnosis of UC up to last follow-up. This study does not require specific procedures as it is intended for the collection and analysis of data from treatments already carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Established diagnosis of UC, defined according to ECCO standard of care
* Documented failure to both anti-TNFα (irrespectively of the number) and vedolizumab
* Ustekinumab or tofacitinib as third-line therapy
* Last follow-up at 24 +/-4 weeks from the start of Ustekinumab or tofacitinib

Exclusion Criteria:

• Patients with unclassified colitis or Crohn disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 100 patients with a diagnosis of UC, defined according to ECCO standard of care and who have been treated with ustekinumab (anti-IL12-23) or tofacitinib (pan JAK inhibitor) and have a follow-up at 24 +/- 4 weeks from the start of the third line therapy. Patients will be enrolled from all the 17 centers participating to this international multicenter study Patients will be managed in each IBD center according to standard of care. All centers will be asked to fill the case report form (CRF) with all patients' data.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Determine which drug between ustekinumab and tofacitinib as a third-line treatment, in cases refractory to both anti-TNFα and vedolizumab, is the best option to achieve disease control in terms of hospitalization rate, surgery rate, drug optimization. | 2 months
  The aim of this retrospective multicentric observational study is to determine which between ustekinumab (anti-IL12-23) and tofacitinib (pan JAK inhibitor) as third-line therapy in UC cases refractory to both anti-TNFα and vedolizumab (inhibitor of α4β7 integrin) is the best compound to achieve disease control.The primary goal is to compare the hospitalization rate, surgery rate, drug optimization rate and the drug discontinuation rate, as a composite primary objective, in patients on either of the two drugs.
  The induction phase of Ustekinumab consists of approximately 6mg/kg intravenous dose administration. After the induction, the maintenance phase consists of a 90mg subcutaneous dose every 8 weeks. The induction phase of Tofacitinib consists of 10mg twice daily for 8 to 16 weeks. After the induction, the maintenance phase consists of 5mg x twice daily.

SECONDARY OUTCOMES:
IBD outcomes | 2 months
  * hospitalization rate (e.g. hospitalization, admission to intensive care unit)
  * surgery rate (type of surgery, occurrence colorectal dysplasia and/or colorectal cancer)
  * drug optimization rate (start of systemic steroids, immunosuppressants, or biologics, dose optimization, interval optimization), switch to another drug, or swap to another drug
  * drug discontinuation rate alone (need to switch or to swap to another drug)

CONTACTS AND LOCATIONS:
Overall Officials: MARIANGELA ALLOCCA, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Mariangela Allocca, Milan, Italy